CLINICAL TRIAL: NCT05094180
Title: Open Label Randomized Clinical Trial to Assess the Safety of Teleconsultation, Compared to the Traditional Clinical Consultation
Brief Title: Open Label Randomized Clinical Trial to Assess the Safety of Teleconsultation
Acronym: ECASeT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSAPG-15
Record Dates: First submitted 2021-10-03; First posted 2021-10-26 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Various Clinical Conditions Commonly Followed up in a Secondary Hospital
MeSH Terms: interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-face consultation (Other)
  Interventions: Other: Face-to-face appointment
- Remote consultation (telephone or video consultation mode) (Active Comparator)
  Interventions: Other: Remote consultation (telephone or video consultation mode)

INTERVENTIONS:
Other: Face-to-face appointment — Participants will be scheduled with face-to-face appointments as usual (control arm). All phone calls (except reminders for scheduled visits) performed by the physician during the study will be recorded. Per protocol, participants allocated in the control arm can receive up to 25% of physician-doctor interactions by phone (that is, one phone call allowed for three face-to-face appointments).
  Arms: Face-to-face consultation
Other: Remote consultation (telephone or video consultation mode) — Patients will be seen through one of the two remote consultation modalities: video consultation or telephone. Patients will receive a reminder by text or call before the appointment.
  In the case of telephone consultation, patients will be informed of the date and time slot in which they must wait for the doctor's call. At the time of the appointment, the doctor will call the contact phone number of the patients and/or their family members, starting with the first contact number that appears in the patient's medical history, and using the rest of the contacts available if there is no response. .
  In the case of video consultation, at the time of the appointment, patients will receive a link to the application that manages the teleconsultation. Once in the application, they will remain in the virtual waiting room until the doctor switches to the videoconference.
  Arms: Remote consultation (telephone or video consultation mode)

SUMMARY:
Randomized-controlled trial to assess the safety of remote consultations (both video and teleconsultation) in the follow-up of patients in the hospital setting. A total of 2136 patients will be randomly allocated into one of the three study arms: A) face-to-face consultation (control) B) Remote consultation (telephone or video consultation). Primary outcome will be the frequency of complications of the underlying disease, including adverse reactions to the treatment of the underlying disease.

To be eligible for remote consultation, patients have to have adequate digital literacy at physician discretion, technological capacity to use the video conferencing software, and undergo a type of follow-up that, due to the moderate complexity of the pathology, do not require physical examinations. Patients followed up in more than three departments, those with visual or hearing impairments that may hamper patient-physician communication, and those enrolled in another clinical trial that requires an experimental intervention during the follow-up will be excluded from the study.

Physicians can schedule and cancel appointments at their discretion. At least three visits should be scheduled in the study setting: the baseline visit (i.e., screening visit), intermediate visits (pre-defined by the physician based on the follow-up needed for managing the baseline condition), and the final visit (i.e., either the follow-up visit closest to 12 ± 2 months after enrollment or before in case of discharge or early discontinuation).

The primary objective will be assessed using a non-inferiority analysis of the cumulative incidence of complications of the baseline disease between remote consultation (video and teleconsultation arms) and face-to-face consultation, using a non-inferiority margin of 2%. The analysis will be based on a modified binomial test to assess the non-inferiority of an experimental intervention vs. a control group in a three-arm trial. The primary analysis will be conducted on a per-protocol study sample, which will include all participants who have finished the study and have not been withdrawn because of non-allowed visits using modalities other than scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of any age.
* Possibility of making consultations by telephone, at the discretion of the investigator, taking into account the severity and complexity of the baseline pathology and the objective of health care.
* Forecast to carry out follow-up in external consultation.
* Agreement to be attended through a non-face-to-face system.
* Ability to connect to the video consultation system.
* Device compatible with the video consultation system.
* Possibility of collaborating in the necessary evaluations.
* Legal capacity to give informed consent.
* Signature of the informed consent for inclusion of the study.

Exclusion Criteria:

* Need to carry out physical examinations, visualize the patient in person or perform techniques that involve face-to-face visits.
* Need for face-to-face consultation due patient's clinical situation.
* Follow-up by more than three medical specialists.
* Visual, hearing or functional impairments that may hamper patient-physician communication.
* Patients enrolled in another clinical trial that requires an experimental intervention during the follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2136 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complications of the underlying disease | 12 months
  Frequency of complications of the underlying disease, including adverse reactions to the treatment of the underlying disease

SECONDARY OUTCOMES:
Severe complications of the baseline disease | 12 months
  Frequency of severe complications of the underlying disease.
Treatment Serious Adverse Event | 12 months
  Frequency of Serious Adverse Events related to the underlying disease's treatment
Avoidable hospitalizations | 12 months
  Total and avoidable hospitalizations, secondary to ambulatory care sensitive conditions
Number of unscheduled medical contacts | 12 months
  Count of unscheduled medical contacts (phone calls, unscheduled visits, ER visits, and admissions) registered in the hospital information system
Care process indicators | 12 months
  Number of consultations made in a format different from the one initially foreseen (face-to-face, telephone consultation or video consultation) Number of empty consultations (the patient does not attend) Number of patients who interrupt their outpatient follow-up Number of prescriptions and type of prescription
Healthcare expenditure | 12 months
  Estimated healthcare expenditure associated with each of the three interventions
Usability of video consultation system | 12 months
  Usability of video consultation system, measured by using the Computer System Usability Questionnaire
Satisfaction of users (health professionals and patients) with the process of clinical care | 12 months
  Degree of satisfaction of users (health professionals and patients) with the process of clinical care, measured by using the satisfaction questionary of the Pla d'enquestes de satisfacció del CatSalut

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Residència Sant Camil, Sant Pere de Ribes, Barcelona
  - Hospital Comarcal de l'Alt Penedès, Vilafranca del Penedès, Barcelona
  - Centre de Rehabilitació, Vilanova i la Geltrú, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez-Molinero A, Carot-Sans G, Escrig R, Tebe C, Arce J, Perez-Lopez C, Ballesta S, Verdejo G, Cedeno A, Riera-Pagespetit M, Vivas-Angeles S, Alarcon JL, Navarro I, Toro S, Mateo L, Torres AJ, Delmas G, Camell H, Chamero A, Gasol M, Piera-Jimenez J; ECASeT Research Group. Study protocol of a randomized controlled trial to assess safety of teleconsultation compared with face-to-face consultation: the ECASeT study. Trials. 2023 Dec 8;24(1):797. doi: 10.1186/s13063-023-07679-1. PMID 38066614